CLINICAL TRIAL: NCT00817817
Title: An Open-Label, Comparative, Randomized, Parallel, Multicenter Study to Determine the Efficacy and Safety of Two Dry Powder Inhalers (DPIs) Used for the Application of Mometasone in the Treatment of Asthma
Brief Title: A Study to Determine the Efficacy and Safety of Two Mometasone Dry Powder Inhalers in the Treatment of Asthma (Study P02524)
Status: Completed | Phase: Phase 3 | Type: Interventional
Sponsor: Organon and Co (Industry)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: None | Purpose: Treatment
Other Study IDs: P02524
Record Dates: First submitted 2009-01-06; First posted 2009-01-07 (Estimated); Last update posted 2024-08-15 (Actual); Status verified 2022-02

CONDITIONS: Asthma
MeSH Terms: conditions — Asthma

STUDY DESIGN:
Oversight: Data Monitoring Committee: No

ARMS (2):
- Group 1 (Experimental)
  Interventions: Device: MF
- Group 2 (Experimental)
  Interventions: Device: MF

INTERVENTIONS:
Device: MF — One evening dose of dry powder inhaled MF 400 μg (Multidose device).
  Other Names: Asmanex; SCH 32088
  Arms: Group 1
Device: MF — One evening dose of dry powder inhaled 400 μg (400 μg capsules - Monodose).
  Other Names: Asmanex; SCH 32088
  Arms: Group 2

SUMMARY:
This is an open-label, comparative, randomized, parallel, multicenter study in asthmatics to determine whether the administration of dry powder inhaled mometasone furoate (MF) 400 μg in a monodose capsule device would be comparable to administration of powder inhaled MF 400 μg in a multidose device.

ELIGIBILITY:
Inclusion Criteria:

* Must be >=18 years of age, of either gender & of any race.
* Must have had a diagnosis of asthma for at least 6 months, characterized by recurrent episode of wheezing, breathlessness, chest tightness & coughing.
* Baseline FEV1 must be >=55% and <=85% of predicted at the Screening Visit, when all restricted medications have been withheld for the specified intervals.
* Must demonstrate evidence of an increase in absolute FEV1 of >=12%, with an absolute volume increase of at least 200 mL, after reversibility testing at the Screening Visit or documented in the patients chart reversibility up to 1 year previous to inclusion.
* Must be free of any clinically significant disease (other than asthma), that would interfere with study evaluations.
* Must be willing to give written informed consent and be able to adhere to dose & visit schedules.
* Must agree to inform their own usual treating physician about their participation in the study.
* Non-pregnant women of childbearing potential must be using a medically acceptable, adequate form of birth control. This includes: 1) hormonal contraceptive as prescribed by a physician (eg, oral combined, hormonal implant, depot injectable); 2) medically prescribed IUD; 3) condom in combination with a spermicide; 4) Monogamous relationship with a male partner who has had a vasectomy or is using a condom plus spermicide during the study. They must have started this birth control method at least 3 months prior to Screening (with the exception of condom in combination with a spermicide), & must agree to continue its use for the duration of the study. Women of childbearing potential who are not currently sexually active must agree and consent to using a double-barrier method should they become sexually active during the course of this study. Women who are surgically sterilized or are at least 1 year postmenopausal are considered not to be of childbearing potential. However, all female subjects must have a urine pregnancy test obtained at screening, prior to initiation of treatment, & at the end of the trial, which must be negative.
* Subjects who did not use the following medication prior to inclusion:

  * Beta 2 agonist short-acting (inhaled, oral)(12 Hours)
  * Beta 2 agonist long-acting (inhaled)(48 Hours)
  * Ipratropium bromide (12 hours)
  * Cromolyn sodium, nedocromil (7 days)
  * Astemizole (3 months)
  * Cetotifeno (3 months)
  * Another investigational drug (1 month)
  * Theophyline (2 weeks)
  * Antihistamines (7 days)
  * Anticholinergics (7 days)
  * Leukotriene modifiers (2 weeks)
  * Oral decongestant long-acting (72 hours)
  * Oral decongestant short-acting (24 hours)
  * Oral corticosteroids (1 month)
  * Injected corticosteroids (3 months)
  * Inhaled corticosteroids (24 hours)
* Baseline portable Peak Expiratory Flow at the Screening Visit must be >50% of predicted. The best value out of 3 must be considered.

Exclusion Criteria:

* Women who are pregnant, breast-feeding, or are pre-menarcheal.
* Have used any investigational drug within the last 30 days or who have ever been treated with any investigational antibody for asthma or rhinitis.
* Are receiving escalating doses of immunotherapy, oral immunotherapy or short course (rush) immunotherapy.
* No subject participating in this study may participate in this same study at another investigational site or in any other investigational study at the same time.
* Must not be randomized into the study more than once.
* Subjects with the following clinical conditions/demography:

  * Allergic to corticosteroids or beta-agonists.
  * Required hospitalization for asthma control within the previous 3 months.
  * Required ventilator support for respiratory failure secondary to their asthma within the last 5 years.
  * Treated in the ER (for a severe asthma exacerbation), or admitted to the hospital for management of airway obstruction, on 2 or more occasions within the last 6 months.
  * Clinical evidence of emphysema, chronic bronchitis, bronchiectasis, or cystic fibrosis.
  * Significant history of renal, hepatic, cardiovascular, metabolic, neurologic, hematological, respiratory, gastrointestinal, cerebrovascular, or other significant medical illness or disorder which, in the judgment of the investigator, could have interfered with the study, or required treatment which might have interfered with the study.
  * Requiring the use of >12 puffs per day of Salbutamol on any 2 consecutive days between study visits.
  * Experienced upper or lower respiratory tract infection within the previous 2 weeks prior to enrollment.
  * Clinically relevant abnormal baseline vital sign.
  * Clinically significant abnormalities on chest x-ray at the Screening Visit or within the previous 6 months.
  * Evidence of clinically significant oropharyngeal candidiasis.
  * Smokers, or ex-smokers who are smoking or have smoked at least 20 years/pack or subjects who are smoking in the last 6 months.
  * Known to be HIV positive.
  * Known to be illicit drug abusers.
  * HPA axis disturbances.
  * Showing any clinical condition considered to be severe.
  * Severe airflow obstruction showing to be life-threatening.
  * Baseline FEV1 <55% of the predicted normal.
  * Uncontrolled hypertension.
  * Suspected pneumonia, pneumothorax, pneumomediastinum, pulmonary TB, alpha-1 anti-trypsin deficiency, lung mycosis or pulmonary cystic fibrosis.
  * History of thoracic surgery or any previous malignancy of the lung,
  * Significant heart disease,
  * Receiving beta-adrenergic blocking agents.
* Presenting baseline portable peak expiratory flow at the Screening Visit <=50% of predicted. The best value out of 3 must be considered.

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 93 (Actual)
Dates: Start 2002-10-01 (Actual); Primary Completion 2003-05-01 (Actual); Study Completion 2003-05-01 (Actual)

PRIMARY OUTCOMES:
The assessment of efficacy will be done by spirometry, determining the difference in FEV1 and PEFR measured by spirometry on baseline, 7, 14, 28, 42 and 56 days after initiation of MF dry powder inhaler (DPI) therapy. | Baseline, 7, 14, 28, 42, and 56 days after initiation of MF DPI therapy.
To determine the number of puffs/day of rescue medication (Salbutamol). | Daily

SECONDARY OUTCOMES:
To compare the PEFR daily measurements obtained by Peak flow Meter used by subjects at home. | Daily
To compare the daily scores for asthma symptoms and sleep quality. | Every morning
To compare the evaluation of response to therapy made by the investigator at each visit compared to the Baseline visit. | Visits 2 to 6.
To determine and compare the safety (HPA axis evaluation) of both treatments using 400 μg MF DPI once daily in adult subjects with asthma. | Visits 2 to 6
To determine and compare the safety (clinical laboratory measurements) of both treatments using 400 μg MF DPI once daily in adult subjects with asthma. | Visit 6
To determine and compare the tolerability (adverse events) of both treatments using 400 μg MF DPI once daily in adult subjects with asthma. | Visits 2 to 6.

REFERENCES:
- [Result] Pereira CA, Vianna FF, Cukier A, Stelmach R, Oliveira JC, Carvalho EV, Gomes EP, Mayo SV, Chibante AM, Domingues CP. Efficacy and safety of two dry-powder inhalers for the administration of mometasone furoate in asthma patients. J Bras Pneumol. 2010 Jul-Aug;36(4):410-6. doi: 10.1590/s1806-37132010000400004. English, Portuguese. PMID 20835586